CLINICAL TRIAL: NCT01796223
Title: Effects of Systematic Patient Feedback on Therapy Outcome and Dropout: A Randomized Controlled Study on Adult Out-patients at a Community Mental Health Centre.
Brief Title: Effects of Systematic Patient Feedback on Therapy Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/1271; 2011/1271 (Registry Identifier: Regional committee for medical research ethics)
Record Dates: First submitted 2013-02-19; First posted 2013-02-21 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Mental Disorders
Keywords: Community mental health services; Psychotherapy; Physician-Patient Relations; Norway
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feedback (Experimental): Feedback system included in psychotherapy
  Interventions: Behavioral: Feedback
- control (Active Comparator): Psychotherapy as usual
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Feedback — The Partners for Change Outcome Management System, administered at the beginning and ending of every therapy session.
  Other Names: PCOMS; KOR (Norwegian)
  Arms: Feedback
Behavioral: Control
  Arms: control

SUMMARY:
The aim of this study is to evaluate the effects of a feedback-system in psychotherapy on adult out-patients at a community mental health centre. It is hypothesized that the intervention will lead to more effective treatment, decreasing treatment dropout as well as improving patient-therapist relationship and patient activation in treatment.

ELIGIBILITY:
The aim is to include a total of 128 patients.

Inclusion Criteria:

* Referred for treatment of mental disorder(s)

Exclusion Criteria:

* Psychiatric emergency
* Poor/no understanding of Norwegian language
* Lack of ability to execute the practical procedures required for the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Health care utilization | 12 months
  Referral- and drop-out rate

SECONDARY OUTCOMES:
Symptom level | T 0 (baseline) and T4 (6 months, end of treatment)
  Outcome Rating Scale and BASIS 32 and WHO-5
Patient satisfaction | T0, T2 (2 months), T4 (6 months, end of treatment)
  Client Satisfaction Questionnaire (CSQ-8; Attkinson & Zwick, 1982)
Level of functioning | T1 (1 hour start of treatment) and T4 (6 months or end of treatment)
  Global Assessment of Functioning (GAF; Hall, 1995)
Preferences for involvement in decision making | T0, T2 (2 months) and T3 (3 months)
  Modified Control Preferences Scale (6 items)
Patient Activation Measure | T0, T1 (1 hour start of treatment), T3 (3 months) and T4 (6 months)
  Patient Activation Measure Mental Health Questionnaire (13 items)
Alliance | T1 (1 hour start of treatment), T2 (2 months
  Working Alliance Inventory (WAI-S)

OTHER OUTCOMES:
Use of health services | 12 months
  Number of visits at general practitioner or other health services

CONTACTS AND LOCATIONS:
Overall Officials: Olav M Linaker, MD, PhD, Study Chair — Norwegian University of Science and Technology; Mariela M Lara, MA, Principal Investigator — National Taiwan Normal University
Locations (1):
- Tiller Distriktspsykiatriske Senter, Trondheim, Norway

REFERENCES:
- [Result] Brattland H, Koksvik JM, Burkeland O, Grawe RW, Klockner C, Linaker OM, Ryum T, Wampold B, Lara-Cabrera ML, Iversen VC. The effects of routine outcome monitoring (ROM) on therapy outcomes in the course of an implementation process: A randomized clinical trial. J Couns Psychol. 2018 Oct;65(5):641-652. doi: 10.1037/cou0000286. Epub 2018 Aug 16. PMID 30113180
- [Derived] Brattland H, Koksvik JM, Burkeland O, Klockner CA, Lara-Cabrera ML, Miller SD, Wampold B, Ryum T, Iversen VC. Does the working alliance mediate the effect of routine outcome monitoring (ROM) and alliance feedback on psychotherapy outcomes? A secondary analysis from a randomized clinical trial. J Couns Psychol. 2019 Mar;66(2):234-246. doi: 10.1037/cou0000320. Epub 2019 Jan 31. PMID 30702322